CLINICAL TRIAL: NCT05134311
Title: Examining the Use of Three Dimensional Ultrasound in the Assessment of Vascular Pathologies
Acronym: 3D-US
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-1292-NHPP
Record Dates: First submitted 2021-11-03; First posted 2021-11-24 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: PAD - Peripheral Arterial Disease; Vascular Diseases; Wounds
MeSH Terms: conditions — Vascular Diseases; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: The primary analysis will compare the proportion of patients readmitted within 30 days of their ultrasound among those who received the 3D ultrasound vs. those who received the 2D ultrasound using a chi-square test. We will also compare the proportion of patients who showed up for their follow-up appointment among those who received the 3D ultrasound vs. those who received the 2D ultrasound using a chi-square test. We will assess for differences in baseline characteristics and factors known to be associated with readmission and compliance with follow-up among the two groups. If warranted, we will adjust for these differences using multivariable regression models.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D-US (Experimental): These subjects will have a 3D rendering of their vascular testing shown to them.
  Interventions: Device: PIUR tUS Imaging System
- Standard US (No Intervention): These subjects will be shown a hand drawn sketch of the results of the vascular testing.

INTERVENTIONS:
Device: PIUR tUS Imaging System — PIUR imaging has developed PIUR Infinity tUS, a 3D freehand tomographic ultrasound system capable of rapid, safe and accurate reconstructive 3D quantifiable vascular imaging.
  Arms: 3D-US

SUMMARY:
The ability to have a visual aid to depict areas of vascular disease that are affecting the patient's health can help in patient comprehension of the problem. This comprehension can lead to better understanding of the issue and increase patient compliance to treatment. The hand drawn sketch produced by the ultrasound technologist provides an inadequate visualization of the vascular insufficiency that is causing the patient's symptoms.

PIUR imaging has developed PIUR Infinity tUS, a 3D freehand tomographic ultrasound system capable of rapid, safe and accurate reconstructive 3D quantifiable vascular imaging. This system will provide a low cost and reproducible imaging solution that will be an effective educational tool for people with vascular disease.

DETAILED DESCRIPTION:
Peripheral arterial disease (PAD) affects approximately 10% of the American population, with 30% to 40% of these patients presenting with claudication symptoms. The prevalence of PAD increases with age and the number of vascular risk factors. More importantly, it is a marker of atherosclerotic disease burden, and is associated with increased mortality from cardiovascular and cerebrovascular causes. There have been recent advances in noninvasive imaging, endovascular approaches for revascularization, and aggressive risk factor management for prevention of cardiac and cerebrovascular complications in PAD.

Ultrasound scanning imaging systems are currently the primary choice for vascular diagnostics. After a standard vascular study, the ultrasound technologist produces a handwritten sketch that highlights various parameters (vessel size and blood flow) throughout the vasculature in question. This sketch is then interpreted by the physician who then assesses and, if need be, performs interventions. This sketch is shown to the patient to better illustrate the vascular insufficiency issues that are affecting the patient. A digital copy of the sketch is also uploaded to the patient portal.

Due to a limited field of action and poor quantification accuracy, patients are often referred for secondary scanning procedures such as computed tomography angiography, magnetic resonance angiography and catheter angiography for more detailed imaging. Referrals delay treatment, expose the patient to potential health risks and pose higher costs to healthcare providers. This can lead to poor patient compliance and avoidable hospital readmissions. This presents a need to improve the rapidity and safety of the diagnosis of vascular conditions in patients to enable rapid treatment of conditions such as peripheral artery disease. There is also a need for cost effective preventative screening and surveillance to enable early intervention, for example, people at high risk of limb amputation.

The PIUR tUS Imaging System has been approved for use in the European Union for over 1 year. Studies performed in Europe have highlighted the system's ability to accurately depict various pathologies in a 3D form. Currently, there is no market equivalent of this technology approved by the FDA for use in the United States. We are conducting this study to determine whether the 3D images created by the device shown to patients can be used as an educational tool to increase patient comprehension of the disease process, compared with the standard of care 2D images. This will be measured in terms of compliance with follow-up appointments and 30-day readmission rates.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years of age or older
* Suspected vascular insufficiency that requires ultrasound evaluation
* Subject is able to sign a consent form
* Scheduled ultrasound testing at the wound center to evaluate vasculature

Exclusion Criteria:

* Younger than 18 years old
* Subject is not scheduled to have ultrasound testing at the wound center
* Subject is unable to or refuses to consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
30 Day re-admission | 30 Days after imaging
  The primary endpoint of the study will be the treatment outcomes for the patients. We will review readmission rates (30 days from the day of the ultrasound) as well as compliance to first follow-up appointment after the ultrasound of interventional cohort. These endpoints will be compared to those of a historical cohort of persons who were treated for similar pathologies in the past.

CONTACTS AND LOCATIONS:
Overall Officials: Alisha Oropallo, MD, Principal Investigator — Northwell Health Comprehensive Wound Healing & Hyperbaric Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rogers S, Carreira J, Phair A, Olech C, Ghosh J, McCollum C. Comparison Between Below Knee Contrast Enhanced Tomographic 3D Ultrasound and CT, MR or Catheter Angiography for Peripheral Artery Imaging. Eur J Vasc Endovasc Surg. 2021 Mar;61(3):440-446. doi: 10.1016/j.ejvs.2020.10.007. Epub 2020 Nov 20. PMID 33229220
- See also: Company website for 3D imaging device — https://piurimaging.com/

DOCUMENTS (2):
  • Study Protocol (2021-02-26): https://cdn.clinicaltrials.gov/large-docs/11/NCT05134311/Prot_000.pdf
  • Informed Consent Form (2021-03-25): https://cdn.clinicaltrials.gov/large-docs/11/NCT05134311/ICF_001.pdf